CLINICAL TRIAL: NCT04701866
Title: Music as a Potential Intervention to Improve Hemodynamic Tolerability of Repetitive Sub-Anesthetic IV Ketamine Infusions in Bipolar and Unipolar Depression: A Pilot Study
Brief Title: Music as an Intervention to Improve Hemodynamic Tolerability of Ketamine in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Réseau québécois sur le suicide, les troubles de l'humeur et les troubles associés (Unknown)
Responsible Party: Principal Investigator, Stéphane Richard-Devantoy, Principal Investigator, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOUGKMT01
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Unipolar Depression; Depression, Bipolar
Keywords: Treatment-Resistant Depression; Ketamine; Music; Hemodynamic Changes
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depressive Disorder; Bipolar Disorder | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator and outcome assessors will be masked throughout the trial. Participants and clinicians administering the ketamine treatments will not be masked, given the nature of the music intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music (Experimental): Music will be provided for participant's six 40 minute IV infusions of 0.5mg/kg ketamine administered over four weeks (biweekly for 2 weeks, then weekly for 2 weeks).
  Interventions: Other: Music
- Usual Care (No Intervention): Participant's six 40 minute IV infusions of 0.5mg/kg ketamine administered over four weeks (biweekly for 2 weeks, then weekly for 2 weeks) will be administered as per usual care. That is, without music provided or permitted. Contact time with clinicians before, during, and after ketamine treatments will be matched.

INTERVENTIONS:
Other: Music — Music will be provided via headphones during all 6 ketamine treatments, beginning at the commencement of each infusion and ending 55 minutes later. On the day of each infusion, before the treatment begins, clinicians will discuss music choices with participants in order to select amongst one of several options that have been designed for this purpose (length, genre, intensity, etc.).
  Arms: Music

SUMMARY:
The purpose of this study is to assess the impact of music on patients receiving a course of intravenous (IV) ketamine for treatment-resistant depression (TRD), both unipolar and bipolar. The primary outcome is changes in in systolic blood pressure throughout each 40-minute infusion. Secondary outcomes include repeated measures of mood, anxiety, suicidality, and psychological/physical pain. Aspects of the treatment experience, with and without music, will also be explored.

DETAILED DESCRIPTION:
Depression is the first cause of disability worldwide, and approximately 1 in 3 patients will fail to respond to current treatments. Intravenous (IV) low-dose ketamine has remarkable efficacy in even the most treatment-resistant depression (here defined as failure to at least two adequate trials of Level 1-evidence psychiatric medications), inducing remission in 25-50%.

Over 100 randomized clinical trials (RCTs) show that music can mitigate hemodynamic and psychological stress caused by even highly invasive medical procedures. Though never studied, music may similarly improve ketamine tolerability.

In this randomized, single-blind (assessors will not know whether participants receive music or not) single-center trial, 20 participants with TRD will receive 1) curated music or 2) no music during their course of 6 IV ketamine treatments (0.50mg/kg bodyweight) over 4 weeks. The primary aim is to compare changes in systolic blood pressure from the beginning to the end (40 minutes, peak plasma concentration) of each infusion between groups.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar and unipolar depressive episode, current episode of depression (DSM-V) despite at least two adequate trials of Level 1-evidence psychiatric medications.
* No active substance use disorder (beyond nicotine use disorder);
* No contraindication of ketamine;
* Not of childbearing potential, defined as: Postmenopausal (defined as no menses for 12 months without an alternative medical cause). A high follicle stimulating hormone (FSH) level (>40 IU/L or mIU/mL in the postmenopausal range) will be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy, however in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient;
* Permanently sterile: permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy.
* Female subjects of childbearing potential must have a negative urine pregnancy test at the beginning and be willing to use a highly effective method of contraception during the treatment and after the last ketamine infusion.
* Female subjects of childbearing potential must practice a highly effective method of contraception (failure rate of <1percent per year when used consistently and correctly) beginning at least two weeks before and continued while receiving ketamine infusions;
* Male subjects who are sexually active with a woman of childbearing potential must agree to use a double-barrier method of contraception (eg, diaphragm or cervical/vault caps plus condom with spermicidal foam/gel/film/cream/suppository).
* Male subjects who are sexually active with a woman who is pregnant must agree to use a condom. Male subjects must also agree to not donate sperm during the treatment and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of ketamine;
* Abstention from consuming grapefruit juice (a potent 3A4 cytochrome inhibitor) on the day of the ketamine infusions as it may alter the metabolism of ketamine;
* Provision of written informed consent after reading the participant information handout;

Exclusion Criteria:

* Baseline blood pressure within normal limits, i.e. below 140/90 mmHg, when measured thrice in a quiet room.
* Significant hearing impairment not improved with hearing aids and/or sound amplification or unwillingness to listen to music during treatment;
* The subject's depressive symptoms have previously demonstrated non-response to esketamine or ketamine in the current major depressive episode;
* Known intellectual deficiency or autism spectrum disorder;
* Unable to accommodate regular visits to the Depressive Disorders Program at the Douglas Mental Health University Institute, Montreal, QC;
* Depression evaluated as secondary to stroke, cancer or other severe medical illnesses;
* Known risk factors for intracranial hemorrhage, including previous significant trauma, known aneurysm, or previous neurosurgery;
* Evidence of clinically relevant disease, e.g., renal or hepatic impairment, significant coronary artery disease (myocardial infarct within a year prior to initial randomization), cerebrovascular disease, viral hepatitis B or C, acquired immunodeficiency syndrome;
* Prior or current substance abuse or dependence (except for caffeine or nicotine dependence) and/or recent history (last 12 months) of alcohol or cannabis abuse or dependence, as defined by DSM-5 criteria. (Cannabis will be considered similarly to alcohol for the purpose of this study, as it is clinically, in the context of its legalization in Canada. That is, recreational use that does not meet criteria for a substance use disorder and/or is not deemed to be negatively impacting participants' physical and mental health will not justify exclusion from the study just as it does not justify exclusion from purely clinical treatment by ketamine.)
* A positive toxicology screen for drugs that are not prescribed;
* Unwilling, or unable to receive treating physician's agreement, or unable to hold benzodiazepines from the evening prior to the infusion of ketamine;
* Unwilling, or unable to receive treating physician's agreement, to discontinue any narcotic beginning a minimum of 5 drug half-lives prior to infusion;
* Unwilling, or unable to receive treating physician's agreement, to discontinue memantine (an NMDA antagonist) during infusions, beginning a minimum of 5 drug half-lives prior to infusions;
* Pregnant, lactating, or of childbearing potential and not willing to use an approved method of contraception during the ketamine infusion, as per above;
* A clinical finding that is unstable or that, in the opinion of the treating clinician(s), would be negatively affected by, or would affect, the medication (e.g., diabetes mellitus, unstable angina);
* Liver function tests AST and ALT three times the upper normal limit at screening.
* Uncorrected hypothyroidism or hyperthyroidism: Subjects needing a thyroid hormone supplement to treat hypothyroidism must have been on a stable dose of the medication for 3 months prior to beginning infusions;
* Clinically significant deviation from the reference range in clinical laboratory test results as judged by the clinician(s);
* ECG results considered significantly abnormal as determined by the clinician(s);
* History of seizure disorder, except febrile convulsions;
* Known history of intolerance or hypersensitivity to ketamine;
* Acute psychotic symptoms, as judged by the initial clinical interview or reported by referring clinicians;
* Any significant, recent, acute decline in exercise tolerance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Changes in Systolic Blood Pressure | From 0 to 40 minutes of each infusion.
  For the primary outcome data analysis, we will adopt the generalized linear model (GLM) to investigate the change in systolic blood pressure (SBP) at 40 minutes versus at 0 minutes between intervention and control groups. Specifically, we treat the difference between the average of the triplicate SBP measurements (measured by a calibrated Welch Allyn Blood Pressure Device at 0 minutes and the average of the triplicate SBP measurements at 40 minutes at each infusion as the outcomes in the GLM, adjusting for covariates such as intervention, age and sex. The generalized estimating equation (GEE) technique is proposed to estimate the regression coefficients, and the corresponding variances are estimated by the sandwich estimators.

SECONDARY OUTCOMES:
Change From Baseline in MADRS Total Score to Last Treatment | Baseline, Day 23
  The Montgomery-Åsberg Depression Rating Scale is a 10-item, clinician-rated scale to rate the severity of the depressive symptoms. Each item is scored from 0 (item's symptoms not present) to 6 (item's symptoms are severe). The total possible score is 60. Higher scores indicate greater severity.
Change From Baseline in MADRS Total Score to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Montgomery-Åsberg Depression Rating Scale is a 10-item, clinician-rated scale to rate the severity of the depressive symptoms. Each item is scored from 0 (item's symptoms not present) to 6 (item's symptoms are severe). The total possible score is 60. Higher scores indicate greater severity.
Change From Baseline in Beck Depression Inventory (BDI-II) Total Score to Last Treatment | Baseline, Day 23
  The Beck Depression Inventory Scale is a 21-item, patient-rated scale to rate the severity of the depressive symptoms. Each item is scored from 0 (item's symptoms not present) to 3 (item's symptoms are severe). The total possible score is 63. Higher scores indicate greater severity.
Change From Baseline in Beck Depression Inventory (BDI-II) Total Score to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Beck Depression Inventory Scale is a 21-item, patient-rated scale to rate the severity of the depressive symptoms. Each item is scored from 0 (item's symptoms not present) to 3 (item's symptoms are severe). The total possible score is 63. Higher scores indicate greater severity.
Change From Baseline in Clinician-Rated Global Impression Improvement Score to Last Treatment | Baseline, Day 23
  The Clinician-Rated Global Impression Improvement score (CGI-I) rates improvement with treatment from 1 to 7, with higher scores indicating a worse outcome.
Change From Baseline in Clinician-Rated Global Impression Severity Score to Last Treatment | Baseline, Day 23
  The Clinician-Rated Global Impression Severity score (CGI-S) rates severity of illness from 1 to 7, with higher scores indicating a worse outcome.
Change From Baseline in Clinician-Rated Global Impression Suicidality Severity Score to Last Treatment | Baseline, Day 23
  The Clinician-Rated Global Impression Suicidality Severity score (CGI-SS) rates severity of suicidality from 1 to 5, with higher scores indicating a worse outcome.
Change From Baseline in Clinician-Rated Global Impression Suicidality Improvement Score to Last Treatment | Baseline, Day 23
  The Clinician-Rated Global Impression Suicidality Improvement score (CGI-SI) rates the improvement in suicidality from 1 to 7, with higher scores indicating a worse outcome.
Change From Baseline in Clinician-Rated Global Impression Improvement Score to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Clinician-Rated Global Impression Improvement score (CGI-I) rates improvement with treatment from 1 to 7, with higher scores indicating a worse outcome.
Change From Baseline in Clinician-Rated Global Impression Severity Score to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Clinician-Rated Global Impression Severity score (CGI-S) rates severity of illness from 1 to 7, with higher scores indicating a worse outcome.
Change From Baseline in Clinician-Rated Global Impression Suicidality Severity Score to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Clinician-Rated Global Impression Suicidality Severity score (CGI-SS) rates severity of suicidality from 1 to 5, with higher scores indicating a worse outcome.
Change From Baseline in Clinician-Rated Global Impression Suicidality Improvement Score to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Clinician-Rated Global Impression Suicidality Improvement score (CGI-SI) rates the improvement in suicidality from 1 to 7, with higher scores indicating a worse outcome.
Change From Baseline in PSQI Total and Subscores to Last Treatment | Baseline, Day 23
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions. The answers refer to the majority of days and nights in the past month. The 19 items are combined to form 7 components, rated from 0 (no difficulty) to 3 (severe difficulty), for a sum of 21 points. A low score indicates better outcome.
Change From Baseline in PSQI Total and Subscores to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions. The answers refer to the majority of days and nights in the past month. The 19 items are combined to form 7 components, rated from 0 (no difficulty) to 3 (severe difficulty), for a sum of 21 points. A low score indicates better outcome.
Change From Baseline in Beck Scale for Suicide Ideation (SSI) Total to Last Treatment | Baseline, Day 23
  The Beck Scale for Suicide Ideation (Current) consists of 19 statements to be rated by the participant on a scale of 0 to 2. A lower score means better outcome.
Change From Baseline in Beck Scale for Suicide Ideation (SSI) Total to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Beck Scale for Suicide Ideation (Current) consists of 19 statements to be rated by the participant on a scale of 0 to 2. A lower score means better outcome.
Change From Baseline in Psychological and Physical Pain to Last Treatment | Baseline, Day 23
  The Visual-Analogue Scales of Psychic and Physical pain consists of two sets of 3 10cm scales. Participants note with a vertical line the intensity of their pain; currently, maximally in the past 15 days, and average over the past 15 days. The left limit indicates "0" pain whereas the right bound indicates "maximal" pain.
Change From Baseline in Psychological and Physical Pain to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The Visual-Analogue Scales of Psychic and Physical pain consists of two sets of 3 10cm scales. Participants note with a vertical line the intensity of their pain; currently, maximally in the past 15 days, and average over the past 15 days. The left limit indicates "0" pain whereas the right bound indicates "maximal" pain.
Change From Baseline in STAI-Y A to Last Treatment | Baseline, Day 23
  The State-Trait Anxiety Scale (STAI-Y A) consists of 20 participant-rated statements, from 1 to 4 (1= Not at all, 4= Very much so) regarding their current anxiety (state). A lower score corresponds to less severity of symptoms.
Change From Baseline in STAI-Y A to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The State-Trait Anxiety Scale (STAI-Y A) consists of 20 participant-rated statements, from 1 to 4 (1= Not at all, 4= Very much so) regarding their current anxiety (state). A lower score corresponds to less severity of symptoms.
Change From Baseline in STAI-Y B to Last Treatment | Baseline, 1-month follow-up (8 weeks)
  The State-Trait Anxiety Scale (STAI-Y B) consists of 20 participant-rated statements, from 1 to 4 (1= Not at all, 4= Very much so) regarding their longstanding anxiety (trait). A lower score corresponds to less severity of symptoms.
Change From Baseline in STAI-Y B to Follow-up | Baseline, 1-month follow-up (8 weeks)
  The State-Trait Anxiety Scale (STAI-Y B) consists of 20 participant-rated statements, from 1 to 4 (1= Not at all, 4= Very much so) regarding their longstanding anxiety (trait). A lower score corresponds to less severity of symptoms.
The Mystical Experience Questionnaire (MEQ) after each treatment | Immediately after the interventions
  The Mystical Experience Questionnaire consists of 30 statements to rate from 0 (none) to 5 (extreme). Possible scores range from 0 to 150 with higher scores indicating greater mystical experiences.
The Psychedelic Music Questionnaire Short-Form (PMQ-SF) after each treatment | Immediately after the interventions
  The Psychedelic Music Questionnaire Short-Form consists of 15 statements rated from 1 (none) to 5 (extremely). Possible scores range from 0 to 75 with higher scores indicating stronger engagement with, and appreciation of, the music experience.
Inflammatory markers before and after the first and last treatment | Treatment 1 and 6 (day 23)
  Blood samples collected from subjects during the first and last treatments, before and after the infusions, totally 4 samples per patient. A panel of inflammatory markers (including interleukin-6, interleukin-1β, interleukin-1ra, interleukin-10, C-reactive protein) will be analyzed to evaluate treatment effects of one and six ketamine infusions in an exploratory fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Richard-Devantoy, MD, PhD, Principal Investigator — Douglas Mental Health University Insitute
Locations (2):
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - Douglas Mental Health University Institute, Montreal, Quebec

REFERENCES:
- [Background] Weinberger AH, Gbedemah M, Martinez AM, Nash D, Galea S, Goodwin RD. Trends in depression prevalence in the USA from 2005 to 2015: widening disparities in vulnerable groups. Psychol Med. 2018 Jun;48(8):1308-1315. doi: 10.1017/S0033291717002781. Epub 2017 Oct 12. PMID 29021005
- [Background] Demyttenaere K, Van Duppen Z. The Impact of (the Concept of) Treatment-Resistant Depression: An Opinion Review. Int J Neuropsychopharmacol. 2019 Feb 1;22(2):85-92. doi: 10.1093/ijnp/pyy052. PMID 29961822
- [Background] Geddes JR, Miklowitz DJ. Treatment of bipolar disorder. Lancet. 2013 May 11;381(9878):1672-82. doi: 10.1016/S0140-6736(13)60857-0. PMID 23663953
- [Background] Pompili M, Gonda X, Serafini G, Innamorati M, Sher L, Amore M, Rihmer Z, Girardi P. Epidemiology of suicide in bipolar disorders: a systematic review of the literature. Bipolar Disord. 2013 Aug;15(5):457-90. doi: 10.1111/bdi.12087. Epub 2013 Jun 12. PMID 23755739
- [Background] Grady SE, Marsh TA, Tenhouse A, Klein K. Ketamine for the treatment of major depressive disorder and bipolar depression: A review of the literature. Ment Health Clin. 2018 Mar 23;7(1):16-23. doi: 10.9740/mhc.2017.01.016. eCollection 2017 Jan. PMID 29955493
- [Background] Fukumoto K, Fogaca MV, Liu RJ, Duman C, Kato T, Li XY, Duman RS. Activity-dependent brain-derived neurotrophic factor signaling is required for the antidepressant actions of (2R,6R)-hydroxynorketamine. Proc Natl Acad Sci U S A. 2019 Jan 2;116(1):297-302. doi: 10.1073/pnas.1814709116. Epub 2018 Dec 17. PMID 30559184
- [Background] De Kock M, Loix S, Lavand'homme P. Ketamine and peripheral inflammation. CNS Neurosci Ther. 2013 Jun;19(6):403-10. doi: 10.1111/cns.12104. Epub 2013 Apr 10. PMID 23574634
- [Background] Chen MH, Li CT, Lin WC, Hong CJ, Tu PC, Bai YM, Cheng CM, Su TP. Rapid inflammation modulation and antidepressant efficacy of a low-dose ketamine infusion in treatment-resistant depression: A randomized, double-blind control study. Psychiatry Res. 2018 Nov;269:207-211. doi: 10.1016/j.psychres.2018.08.078. Epub 2018 Aug 21. PMID 30153598
- [Background] Wan LB, Levitch CF, Perez AM, Brallier JW, Iosifescu DV, Chang LC, Foulkes A, Mathew SJ, Charney DS, Murrough JW. Ketamine safety and tolerability in clinical trials for treatment-resistant depression. J Clin Psychiatry. 2015 Mar;76(3):247-52. doi: 10.4088/JCP.13m08852. PMID 25271445
- [Background] van Schalkwyk GI, Wilkinson ST, Davidson L, Silverman WK, Sanacora G. Acute psychoactive effects of intravenous ketamine during treatment of mood disorders: Analysis of the Clinician Administered Dissociative State Scale. J Affect Disord. 2018 Feb;227:11-16. doi: 10.1016/j.jad.2017.09.023. Epub 2017 Sep 28. PMID 29045915
- [Background] Conrad C, Niess H, Jauch KW, Bruns CJ, Hartl W, Welker L. Overture for growth hormone: requiem for interleukin-6? Crit Care Med. 2007 Dec;35(12):2709-13. doi: 10.1097/01.ccm.0000291648.99043.b9. PMID 18074473
- [Background] Wiwatwongwana D, Vichitvejpaisal P, Thaikruea L, Klaphajone J, Tantong A, Wiwatwongwana A; Medscape. The effect of music with and without binaural beat audio on operative anxiety in patients undergoing cataract surgery: a randomized controlled trial. Eye (Lond). 2016 Nov;30(11):1407-1414. doi: 10.1038/eye.2016.160. Epub 2016 Oct 14. PMID 27740618
- [Background] Merakou K, Varouxi G, Barbouni A, Antoniadou E, Karageorgos G, Theodoridis D, Koutsouri A, Kourea-Kremastinou J. Blood Pressure and Heart Rate Alterations through Music in Patients Undergoing Cataract Surgery in Greece. Ophthalmol Eye Dis. 2015 Jun 11;7:7-12. doi: 10.4137/OED.S20960. eCollection 2015. PMID 26106264
- [Background] Bradt J, Dileo C. Music interventions for mechanically ventilated patients. Cochrane Database Syst Rev. 2014;2014(12):CD006902. doi: 10.1002/14651858.CD006902.pub3. Epub 2014 Dec 9. PMID 25490233
- [Background] Metcalf CS, Huntsman M, Garcia G, Kochanski AK, Chikinda M, Watanabe E, Underwood T, Vanegas F, Smith MD, White HS, Bulaj G. Music-Enhanced Analgesia and Antiseizure Activities in Animal Models of Pain and Epilepsy: Toward Preclinical Studies Supporting Development of Digital Therapeutics and Their Combinations With Pharmaceutical Drugs. Front Neurol. 2019 Mar 27;10:277. doi: 10.3389/fneur.2019.00277. eCollection 2019. PMID 30972009
- [Background] Kaelen M, Barrett FS, Roseman L, Lorenz R, Family N, Bolstridge M, Curran HV, Feilding A, Nutt DJ, Carhart-Harris RL. LSD enhances the emotional response to music. Psychopharmacology (Berl). 2015 Oct;232(19):3607-14. doi: 10.1007/s00213-015-4014-y. Epub 2015 Aug 11. PMID 26257162
- [Background] Kaelen M, Giribaldi B, Raine J, Evans L, Timmermann C, Rodriguez N, Roseman L, Feilding A, Nutt D, Carhart-Harris R. Correction to: The hidden therapist: evidence for a central role of music in psychedelic therapy. Psychopharmacology (Berl). 2018 May;235(5):1623. doi: 10.1007/s00213-018-4886-8. PMID 29582103
- [Background] Fries GR, Walss-Bass C, Bauer ME, Teixeira AL. Revisiting inflammation in bipolar disorder. Pharmacol Biochem Behav. 2019 Feb;177:12-19. doi: 10.1016/j.pbb.2018.12.006. Epub 2018 Dec 24. PMID 30586559
- [Background] Dakwar E, Anerella C, Hart CL, Levin FR, Mathew SJ, Nunes EV. Therapeutic infusions of ketamine: do the psychoactive effects matter? Drug Alcohol Depend. 2014 Mar 1;136:153-7. doi: 10.1016/j.drugalcdep.2013.12.019. Epub 2014 Jan 15. PMID 24480515
- [Background] Niciu MJ, Shovestul BJ, Jaso BA, Farmer C, Luckenbaugh DA, Brutsche NE, Park LT, Ballard ED, Zarate CA Jr. Features of dissociation differentially predict antidepressant response to ketamine in treatment-resistant depression. J Affect Disord. 2018 May;232:310-315. doi: 10.1016/j.jad.2018.02.049. Epub 2018 Feb 17. PMID 29501990
- [Background] Yatham LN, Kennedy SH, Parikh SV, Schaffer A, Bond DJ, Frey BN, Sharma V, Goldstein BI, Rej S, Beaulieu S, Alda M, MacQueen G, Milev RV, Ravindran A, O'Donovan C, McIntosh D, Lam RW, Vazquez G, Kapczinski F, McIntyre RS, Kozicky J, Kanba S, Lafer B, Suppes T, Calabrese JR, Vieta E, Malhi G, Post RM, Berk M. Canadian Network for Mood and Anxiety Treatments (CANMAT) and International Society for Bipolar Disorders (ISBD) 2018 guidelines for the management of patients with bipolar disorder. Bipolar Disord. 2018 Mar;20(2):97-170. doi: 10.1111/bdi.12609. Epub 2018 Mar 14. PMID 29536616
- [Background] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528
- [Background] Glue P, Neehoff S, Sabadel A, Broughton L, Le Nedelec M, Shadli S, McNaughton N, Medlicott NJ. Effects of ketamine in patients with treatment-refractory generalized anxiety and social anxiety disorders: Exploratory double-blind psychoactive-controlled replication study. J Psychopharmacol. 2020 Mar;34(3):267-272. doi: 10.1177/0269881119874457. Epub 2019 Sep 17. PMID 31526207
- [Derived] Greenway KT, Garel N, Dinh-Williams LL, Beaulieu S, Turecki G, Rej S, Richard-Devantoy S. Music as an Intervention to Improve the Hemodynamic Response of Ketamine in Depression: A Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2354719. doi: 10.1001/jamanetworkopen.2023.54719. PMID 38315489
- [Derived] Garel N, Thibault Levesque J, Sandra DA, Lessard-Wajcer J, Solomonova E, Lifshitz M, Richard-Devantoy S, Greenway KT. Imprinting: expanding the extra-pharmacological model of psychedelic drug action to incorporate delayed influences of sets and settings. Front Hum Neurosci. 2023 Jul 18;17:1200393. doi: 10.3389/fnhum.2023.1200393. eCollection 2023. PMID 37533588